CLINICAL TRIAL: NCT06509373
Title: A Portal-based Advance Care Planning Intervention Among Community-Dwelling Persons Living With Cognitive Impairment
Acronym: Portal-Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00112143; 5K23AG070234-03 (NIH)
Record Dates: First submitted 2024-07-12; First posted 2024-07-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Care Planning
Keywords: Advance Care Planning; Mild Cognitive Impairment; Dementia; Patient Portal
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Standard of Care; Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACPVoice Intervention (Experimental): Community-dwelling persons living with cognitive impairment aged 65 and older with known or probable mild cognitive impairment or dementia or elevated eRADAR score (with decision-making capacity), who are affiliated with the Atrium-Wake Forest Baptist Health , have a primary care physician at one of the participating sites, and have an active patient portal account.
  Interventions: Behavioral: Advance Care Planning Tool - ACPVoice
- Standard of Care (Active Comparator): Community-dwelling persons living with cognitive impairment aged 65 and older with known or probable mild cognitive impairment or dementia or elevated eRADAR score (with decision-making capacity), who are affiliated with the Atrium-Wake Forest Baptist Health, have a primary care physician within the Atrium-Wake Forest Baptist Health Network, and have an active patient portal account.
  Interventions: Behavioral: Standard of Care for Advance Care Planning

INTERVENTIONS:
Behavioral: Advance Care Planning Tool - ACPVoice — Eligible patients will be sent a secure MyChart message with a motivational message asking them to complete the advance care planning tool (ACPVoice) with their care partner/surrogate decision-maker or loved one before their upcoming primary care visit. The ACPVoice tool will be attached electronically to the mychart message. A reminder message will be sent to an non-responders with a different motivational message.
  Arms: ACPVoice Intervention
Behavioral: Standard of Care for Advance Care Planning — Patients will have access to the standardized advance care planning questionnaires readily available already within their mychart account which is part of standard of care.
  Arms: Standard of Care

SUMMARY:
The purpose of this research is to examine the feasibility of using a patient portal based advance care planning (ACP) tool to improve ACP discussions and documentation in persons living with cognitive impairment in outpatient primary care.

DETAILED DESCRIPTION:
The goal of this study is to explore whether sending a portal-based ACP tool (called ACPVoice) paired with a motivational message within the patient portal before a routine primary care physician visit can improve ACP discussions and documentation within the electronic health record among persons living with cognitive impairment in outpatient primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years old and older
* Diagnosis of recognized or probable mild cognitive impairment or mild dementia or elevated eRADAR score
* Completed visit with their primary care provider (PCP) within the past 12 months and have upcoming PCP visit in next 6 months
* Have an active patient portal account

Exclusion Criteria:

* Lives in a long-term care facility
* Severe vision impairment/blindness (as they need to be able to read portal messages)
* Enrolled in hospice
* Lacks decisional capacity as deemed by PCP

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Reach/Engagement | 6 months post intervention
  Percentage of participants who open the advance care planning tool (ACPVoice) mychart message
Intervention Completion | 6 months post intervention
  Percentage of participants who were sent the ACPVoice mychart message that complete the ACPVoice tool.

SECONDARY OUTCOMES:
Advance Care Planning Documentation Rates by Primary Care Providers | 12 months pre intervention
  Documentation of advance care planning within the electronic health record by primary care provider.
Advance Care Planning Documentation Rates by Primary Care Providers | 6 months post intervention
  Documentation of advance care planning within the electronic health record by primary care provider.
Advance Care Planning Billing Code Usage | 12 months pre intervention
  Advance care planning billing codes usages will be recorded.
Advance Care Planning Billing Code Usage | 6 months post intervention
  Advance care planning billing codes usages will be recorded.
Documented Designated Surrogate Decision Maker | 12 months pre intervention
  Measured by number of designated surrogate decision makers documented in the electronic health record.
Documented Designated Surrogate Decision Maker | 6 months post intervention
  Measured by number of designated surrogate decision makers documented in the electronic health record.

OTHER OUTCOMES:
Barrier to Adoption | 6 months during the implementation period and up to 6 months post the implementation period
  Data will be collected via qualitative interviews with participants and providers.
Quality of Advance Care Planning Documentation | 6 months during the implementation period and up to 6 months post the implementation period
  High-quality advance care planning documentation will be defined as addressing ≥4 of the 8 core components with 1 point assigned for each of the following questions related to: health-related goals, what matters most/most important in their life, health-related worries/concerns, named surrogate decision-maker, how much information they would like to know, unacceptable states at the end-of-life, goals if their health was to worsen, and questions about advance care planning forms. Score of 0-8 with 0 indicating no advance care planning questions answered to 8 indicating eight core advance care planning questions answered.
Participant Confidence related to PCP knowing what is important to them | 6 months during the implementation period and up to 6 months post the implementation period
  Data will be collected via a RedCap survey asking 5 questions: i. How confident are you your primary care clinician/team knows what is important to you?, ii. How confident are you that what is important to you will determine the medical care you receive in the future? , iii. To what extent did completing this care planning tool increase or decrease your sense of control over medical decisions?, iv. Before completing the care planning tool, did your primary care clinician/team ask what is important to you? , and v. After completing the care planning tool, did your primary care clinician/team ask what is important to you? .
Feeling Heard and Understood | 6 months during the implementation period and up to 6 months post the implementation period
  Data will be assessed via a RedCap survey with 4 questions: I felt heard and understood by this provider and team, I felt this provider and team put my best interests first when making recommendations about my care, I felt this provider and team saw me as a person, not just someone with a medical problem, I felt this provider and team understood what is important to me in my life.
Digital Health Literacy | 6 months during the implementation period and up to 6 months post the implementation period
  Data will be measured using the Brief Digital Health Care Literacy Scale.
Telephone Advance Care Planning Completion Rates | 6 months during the implementation period and up to 6 months post the implementation period
  Defined as the number of patients who complete the advance care planning tool (ACPVoice) over the telephone.
Paper Advance Care Planning Documentation Rates | 6 months during the implementation period and up to 6 months post the implementation period
  Defined as the number of patients who were mailed and completed the advance care planning tool (ACPVoice) via mail.
Preference-concordant care | 6 months during the implementation period and up to 6 months post the implementation period
  Data will be collected via Redcap survey asking "How strongly do you agree or disagree that your current medical/treatment plan meets your preferences".
Provider Survey Score | 6 months post implementation period
  17 multiple choice items regarding provider opinion on the interventions acceptability, appropriateness, feasibility and overall satisfaction. Total score range is 17-84 with a higher score indicating a more favorable opinion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gabbard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No